CLINICAL TRIAL: NCT06227845
Title: Preterm Infant Intestinal Microbiota Development and Maternal Fecal Transplant
Acronym: PREFLOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Helve (Other)
Collaborators: Karolinska Institutet (Other); University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Otto Helve, Docent, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUS/1978/2023
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Microbial Colonization
Keywords: Premature infant; Fecal microbiota transplant; Cesarean section; Immune system development
MeSH Terms: conditions — Communicable Diseases; Premature Birth | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): 10 infants born by CS to screening negative mothers receive an oral maternal fecal transplant (from their own mother) containing 0.35mg/kg of maternal fecal content at the age of 2-7 days of age.
  Interventions: Other: Fecal microbiota transplant
- Control (No Intervention): 12 infants born by CS (8 to screening negative mothers and 4 to screening positive mothers in case of Blastocystis hominis or Dientamoeba fragilis).
- Comparison (No Intervention): Infants born vaginally to mothers with screening negative or mild pathogene findings (Blastocystis hominis or Dientamoeba fragilis)

INTERVENTIONS:
Other: Fecal microbiota transplant — 0.1-0.3 ml liquid containing 3.5 mg/ml of maternal fecal content, (0.35mg/kg)
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to study if a oral maternal fecal transplant given to a premature infant born by cesarean section (CS) is safe. The investigators will also compare the gut microbiome of the infants to those born by CS and not received the transplant and to premature infants born vaginally.

DETAILED DESCRIPTION:
At the Department of Obstetrics at Helsinki University Hospital the investigators will recruit 36 pregnant women (allowing for screening positivity) between 29 and 34 weeks of pregnancy with for example pre-eclampsia or cervix insufficiency, but are otherwise healthy. The mothers fecal sample is carefully screened in case of contagious diseases. The investigators are aiming to recruit 18 mothers with negative screening samples.

The infants are born at gestational week 30-35 either vaginally or by CS. Group A (study group): 10 preterm infants born by CS. These infants will receive a maternal FMT, which will be administered when they tolerate milk at least 40 mL/day. Group B (comparison group): 8 preterm infants from the screening negative mothers and 4 infants from the mothers who have a positive finding in the screening samples (in case the positive finding is a mild pathogen e.g. Dientamoeba fragilis or Blastocystis hominis) born by CS. In case of antibiotic treatment of the infant, the transplant is given not earlier than 48 hours after the last dose, but not later than 7 days of age. Group C: Comparison group of preterm infants born vaginally 30-35 weeks of gestation. For the comparison group, only fecal samples are obtained as in the other groups.

For group A, blood samples are taken on the day of transplant and 1 and 3 days after. The samples are the same as in SECFLOR main trial: research samples and assessment of routine inflammatory markers (such as CBC and CRP).

From the comparison group (B) CRP and blood count samples are taken as ordered by the treating physician. To assess immunological markers a sample of 1 mL is taken at the age of 5-7 days concomitantly with blood samples ordered by the treating physician. No additional samples are taken from the vaginal delivery group.

From all groups: Meconium sample is collected, and then a stool sample on the day of the transplant, and two days after (from the intervention group only) and starting from 1 weeks of age weekly until the age of 4 weeks or until discharged from the intensive unit. After discharge the parents will collect a stool sample of the child at the age of 3, 6, 9 and 12 months.

Blood samples 1-3mL from all infants born by CS (group A and B) are taken at the age of three and six months to assess immunodevelopment.

Methods Fecal samples: The mothers are asked to provide a fresh stool sample at 29-34 weeks. This is processed for DNA isolation and stored in saline and glycerol. A home sampling stool kit is provided for sampling the mothers and infant's feces from diapers. The intestinal microbiota of mothers and infants is determined using 16S rRNA based analysis using next generation sequencing. Fecal DNA is extracted by repeated bead beating and processed for sequencing using pre-defined primers. DNA extractions and MiSeq runs include internal reference samples and a mock community. Metagenomic analysis will be conducted essentially. Resistance genes will be characterized by mapping metagenomic reads nucleotide to nucleotide against the CARD and Resfinder databases to search for acquired antibiotic resistance genes (ARGs).

Blood samples: The development of all major immune cell populations is analyzed by mass cytometry and 267 plasma proteins by immunoassays. About 100 ul whole blood is collected for mass cytometry analysis and mixed with Cytodelics Whole Blood Cell Stabilizer at a ratio of 1:1, incubated in room temperature for 10 minutes and transferred to a 80C freezer for long-term storage awaiting analysis. Plasma samples are obtained, PBMCs are isolated using density gradient-based separation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with preeclampsia or other risk factors of preterm labor (eg cervix insufficiency or placenta previa) between 29+0 - 34+0 weeks of pregnancy.
* Either parent fluent in Finnish.

Exclusion Criteria:

* Women with other significant medical conditions including acute infection, IBD, celiac disease.
* Travelling outside the EU and use of antibiotics during the last 3 months.
* Gestational diabetes with insulin medication.
* Pregnant with multiples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety; Incidence of Treatment- Adverse Events eg. infections and increased need for respiratory support | 3 months
  The primary outcome of the study is safety of the transplantation process. The patients are followed with measurements of markers of inflammation (C-reactive protein (CRP) and blood leucocytes) on the day of transplant and three consecutive days. Clinical symptoms of infection are monitored (such as apnea, tachycardia, fever) as well as symptoms of the gastrointestinal tract (vomiting, diarrhea, feeding intolerance). Any suspected adverse events (such as infections, increased need for respiratory support) are recorded.

SECONDARY OUTCOMES:
The secondary outcome is the difference in heterogeneity of the intestinal microbiome between infants receiving transplant and the control subjects at 3 and 6 months of age. | 6 months
  The investigators focus on the diversity, richness, taxonomic diversity, and transfer of specific bacteria from the mother to the newborn.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Helve, Docent, Principal Investigator — University of Helsinki
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpen N, Brodin P, de Vos WM, Salonen A, Kolho KL, Andersson S, Helve O. Transplantation of maternal intestinal flora to the newborn after elective cesarean section (SECFLOR): study protocol for a double blinded randomized controlled trial. BMC Pediatr. 2022 Sep 29;22(1):565. doi: 10.1186/s12887-022-03609-3. PMID 36175995
- [Background] Korpela K, de Vos WM. Early life colonization of the human gut: microbes matter everywhere. Curr Opin Microbiol. 2018 Aug;44:70-78. doi: 10.1016/j.mib.2018.06.003. Epub 2018 Aug 4. PMID 30086431
- [Background] Van Belkum M, Mendoza Alvarez L, Neu J. Preterm neonatal immunology at the intestinal interface. Cell Mol Life Sci. 2020 Apr;77(7):1209-1227. doi: 10.1007/s00018-019-03316-w. Epub 2019 Oct 1. PMID 31576423
- [Background] Olin A, Henckel E, Chen Y, Lakshmikanth T, Pou C, Mikes J, Gustafsson A, Bernhardsson AK, Zhang C, Bohlin K, Brodin P. Stereotypic Immune System Development in Newborn Children. Cell. 2018 Aug 23;174(5):1277-1292.e14. doi: 10.1016/j.cell.2018.06.045. PMID 30142345
- [Background] Forsgren M, Isolauri E, Salminen S, Rautava S. Late preterm birth has direct and indirect effects on infant gut microbiota development during the first six months of life. Acta Paediatr. 2017 Jul;106(7):1103-1109. doi: 10.1111/apa.13837. Epub 2017 Apr 24. PMID 28316118
- [Result] Korpela K, Helve O, Kolho KL, Saisto T, Skogberg K, Dikareva E, Stefanovic V, Salonen A, Andersson S, de Vos WM. Maternal Fecal Microbiota Transplantation in Cesarean-Born Infants Rapidly Restores Normal Gut Microbial Development: A Proof-of-Concept Study. Cell. 2020 Oct 15;183(2):324-334.e5. doi: 10.1016/j.cell.2020.08.047. Epub 2020 Oct 1. PMID 33007265